CLINICAL TRIAL: NCT02402075
Title: Spinal Motor Evoked Potentials During Neurosurgical Procedures Within the Central Region
Brief Title: Spinal Motor Evoked Potentials in Brain Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Heinrich-Heine University, Duesseldorf (Other)
Collaborators: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Andrea Szelenyi, Professor, Heinrich-Heine University, Duesseldorf
Other Study IDs: ASze_DF_001
Record Dates: First submitted 2015-03-17; First posted 2015-03-30 (Estimated); Last update posted 2015-03-30 (Estimated); Status verified 2015-03

CONDITIONS: Brain Tumor; Glioma
Keywords: muscle motor evoked potentials; spinal motor evoked potentials; D-wave; brain tumor surgery; intraoperative neuromonitoring
MeSH Terms: conditions — Brain Neoplasms; Glioma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Brain tumor: patients with glioma

SUMMARY:
During neurosurgical resection of brain tumors within brain areas for motor control, it is important to monitor motor function. For this muscle motor evoked potentials are used. Those are elicited by transcranial and direct cortical stimulation. Motor responses are recorded from muscles. In neurosurgical procedures for spinal cord tumors, the same methods are used, but additionally motor activity is recorded from the spinal cord. This is called spinal motor evoked potentials. It is known that the relation between spinal and muscle motor evoked potentials helps to extent the resection of spinal cord tumors. This study implements the spinal motor evoked potential into brain tumor surgery and analyses the relationship between spinal and muscle motor evoked potentials. With this, detection of injury to the brain area for motor control might be discovered earlier and thus tumor resection can be performed safely.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* tumor location adjacent to the motor cortex and corticospinal tract

Exclusion Criteria:

* minor
* neurological degenerative diseases
* neurological immunological diseases
* drug abuse
* implanted medical devices such as cardiac pacemaker
* spine deformation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with glioma
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
D-wave measurement | 24 hours
  numeric assessment, amplitude and latency of D-wave
Clinical motor status according to the MRC scheme | 6 months
  clinical motor status according to the MRC scheme

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Szelenyi, MD PhD, Principal Investigator — Neurosurgical Department, Heinrich Heine University
Locations (2):
- Germany (2):
  - Neurosurgical Department, Düsseldorf
  - Department of Neurosurgery, Frankfurt